CLINICAL TRIAL: NCT00740896
Title: Acute Effects of Smoking on Airway Dendritic Cells
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Rostock (Other)
Collaborators: German Research Foundation (Other)
Responsible Party: PD Dr. med. Marek Lommatzsch, University of Rostock
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: LO-2222
Record Dates: First submitted 2008-08-22; First posted 2008-08-25 (Estimated); Last update posted 2009-04-08 (Estimated); Status verified 2009-04

CONDITIONS: Tobacco Use Disorder
Keywords: Cigarette Smoking; Airway dendritic cells
MeSH Terms: conditions — Tobacco Use Disorder; Cigarette Smoking | interventions — Smoking Devices

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Active Comparator): Participants smoke 8 cigarettes in 4 hours.
  Interventions: Behavioral: Smoking
- 2 (Sham Comparator): Participants are not allowed to smoke for 4 hours.
  Interventions: Behavioral: Smoking

INTERVENTIONS:
Behavioral: Smoking — Active Comparator: Participants smoke 8 cigarettes in 4 hours.
  Arms: 1
Behavioral: Smoking — Sham Comparator: Participants are not allowed to smoke for 4 hours.
  Arms: 2

SUMMARY:
Airway dendritic cells control pulmonary immune responses to inhaled particles. It is the aim of the present study to investigate the acute effects of smoking on the number and surface molecule expression of human airway dendritic cells.

ELIGIBILITY:
Inclusion Criteria:

* Active smoking (at least 10 cigarettes per day)
* Age > 18 years

Exclusion Criteria:

* Any chronic diseases
* Any regular medication
* Any signs or symptoms of an acute infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2008-06; Primary Completion 2008-11 (Actual); Study Completion 2008-12 (Actual)

PRIMARY OUTCOMES:
Total number of dendritic cells in bronchoalveolar lavage fluid | June - September 2008

SECONDARY OUTCOMES:
Surface molecule expression on dendritic cells in bronchoalveolar lavage fluid | June - September 2008

CONTACTS AND LOCATIONS:
Overall Officials: Johann C. Virchow, Professor, MD, FRCP, FCCP, Study Chair — University of Rostock
Locations (1):
- University of Rostock, Rostock, Germany

REFERENCES:
- [Background] Bratke K, Klug M, Bier A, Julius P, Kuepper M, Virchow JC, Lommatzsch M. Function-associated surface molecules on airway dendritic cells in cigarette smokers. Am J Respir Cell Mol Biol. 2008 Jun;38(6):655-60. doi: 10.1165/rcmb.2007-0400OC. Epub 2008 Jan 18. PMID 18203971